CLINICAL TRIAL: NCT01510769
Title: A Phase 3 Randomized, Double-Blind, Multicenter, Placebo- Controlled, Combination Study to Evaluate the Efficacy and Safety of Lesinurad and Febuxostat Compared to Febuxostat Alone at Lowering Serum Uric Acid and Resolving Tophi in Subjects With Tophaceous Gout
Brief Title: Combination Treatment Study in Subjects With Tophaceous Gout With Lesinurad and Febuxostat
Acronym: CRYSTAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RDEA594-304; 2011-003768-55 (EudraCT Number)
Record Dates: First submitted 2012-01-12; First posted 2012-01-16 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Tophaceous Gout
MeSH Terms: interventions — lesinurad; Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- lesinurad 400 mg + febuxostat 80 mg (Experimental)
  Interventions: Drug: Lesinurad; Drug: Febuxostat
- lesinurad 200 mg + febuxostat 80 mg (Experimental)
  Interventions: Drug: Lesinurad; Drug: Febuxostat
- placebo + febuxostat 80 mg (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Febuxostat

INTERVENTIONS:
Drug: Lesinurad — Tablets, 400 mg once daily (QD)
  Arms: lesinurad 400 mg + febuxostat 80 mg
Drug: Lesinurad — Tablets, 200 mg QD
  Arms: lesinurad 200 mg + febuxostat 80 mg
Drug: Placebo — Tablets, Placebo QD
  Arms: placebo + febuxostat 80 mg
Drug: Febuxostat — 80 mg

SUMMARY:
This study will compare the serum uric acid lowering effects, clinical benefits, and safety of lesinurad in combination with febuxostat to febuxostat alone in patients with tophaceaous gout.

DETAILED DESCRIPTION:
Febuxostat is an XO (Xanthine Oxidase) Inhibitor approved Urate Lowering Therapy (ULT) for patients with gout. Although febuxostat has been demonstrated to be superior to allopurinol in lowering serum urate (sUA) to < 6mg/dL in 3 randomized, controlled clinical trials, proportions of subjects experiencing a reduction in tophus area and gout flares were not significantly different compared to allopurinol. Although this study will allow subjects who are naïve to ULT to enroll, it is anticipated that the majority of subjects will currently be taking or have previously experienced XO Inhibitor therapy. This trial will enroll a population of subjects with high uric acid body burden, as all must demonstrate the presence of tophi.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the study procedures, the risks involved and willing to provide written informed consent before the first study related activity.
* Subject is willing to adhere to the visit/protocol schedules.
* Subject meets the diagnosis of gout as per the American Rheumatism Association
* Criteria for the Classification of Acute Arthritis of Primary Gout.
* Subject meets one of the following criteria:
* Subjects who are not currently taking an approved ULT must have an sUA value of ≥ 8 mg/dL (476 µmol/L).
* Subjects entering the study on a medically appropriate dose of febuxostat or allopurinol must have an sUA value of ≥ 6.0 mg/dL (357 µmol/L).
* Subject must be able to take gout flare prophylaxis with colchicine or non-steroidal anti-inflammatory drug (NSAID) (including Cox-2 selective NSAID) ± PPI.
* Subject with at least 1 measurable tophus on the hands/wrists and/or feet/ankles ≥ 5 mm and ≤ 20 mm in the longest diameter.
* Body mass index (BMI) < 45 kg/m2

Exclusion Criteria:

* Subject with known hypersensitivity or allergy to febuxostat.
* Subject who is taking any approved urate-lowering medication other than allopurinol or febuxostat that is indicated for the treatment of gout within 8 weeks of the Screening Visit.
* Subject who previously received pegloticase.
* Subject who consumes more than 14 drinks of alcohol per week (eg, 1 drink = 5 oz [150 mL] of wine, 12 oz [360 mL] of beer, or 1.5 oz [45 mL] of hard liquor).
* Subject with a history or suspicion of drug abuse within the past 5 years.
* Subject with a history of myositis/myopathy or rhabdomyolysis.
* Subject that requires or may require systemic immunosuppressive or immunomodulatory treatment.
* Subject with known or suspected human immunodeficiency virus (HIV) infection.
* Subject with a positive test for active hepatitis B or hepatitis C infection.
* Subject with a history of malignancy within the previous 5 years with the exception of non-melanoma skin cancer that has been treated with no evidence of recurrence, treated cervical dysplasia or treated in situ Grade 1 cervical cancer.
* Subject within the last 12 months with: unstable angina, New York Heart Association thrombosis; or subjects currently receiving anticoagulants.
* Subject with uncontrolled hypertension.
* Subject with an estimated creatinine clearance < 30 mL/min.
* Subjects with a creatine kinase > 2.5 x ULN at any time during the Screening Period.
* Subject with active peptic ulcer disease requiring treatment.
* Subject with a history of xanthinuria, active liver disease, or hepatic dysfunction.
* Subject receiving chronic treatment with more than 325 mg of salicylates per day.
* Subject taking valpromide, progabide, or valproic acid.
* Subject who has received an investigational therapy within 8 weeks or 5 half-lives (whichever is longer) prior to the Screening Visit.
* Subject with any other medical or psychological condition, which in the opinion of the Investigator and/or Medical Monitor, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements, or to complete the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Storgard, MD, Study Director — Ardea Biosciences, Inc.
Locations (111):
- United States (88):
  - Birmingham, Alabama
  - Goodyear, Arizona
  - Peoria, Arizona
  - Pheonix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Glendale, California
  - Huntington Beach, California
  - Irvine, California
  - La Jolla, California
  - Los Angeles, California
  - Rancho Cucamonga, California
  - San Diego, California
  - Denver, Colorado
  - Englewood, Colorado
  - Trumball, Connecticut
  - Washington D.C., District of Columbia
  - Boynton Beach, Florida
  - Brooksville, Florida
  - East Brandenton, Florida
  - Fleming Island, Florida
  - Miami, Florida
  - Napels, Florida
  - Pembroke Pines, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Winter Haven, Florida
  - Conyers, Georgia
  - Johns Creek, Georgia
  - Newnan, Georgia
  - Savannah, Georgia
  - Honolulu, Hawaii
  - Meridian, Idaho
  - Chicago, Illinois
  - Gurnee, Illinois
  - Springfield, Illinois
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Frederick, Maryland
  - Kalamazoo, Michigan
  - Southfield, Michigan
  - Jackson, Mississippi
  - Olive Branch, Mississippi
  - Jefferson City, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Mineola, New York
  - New York, New York
  - Calabash, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Columbus, Ohio
  - Middleburg, Ohio
  - Wadsworth, Ohio
  - Oklahoma City, Oklahoma
  - Belle Vernon, Pennsylvania
  - Clairton, Pennsylvania
  - Duncansville, Pennsylvania
  - Jenkintown, Pennsylvania
  - Lansdale, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Scottdale, Pennsylvania
  - Sellersville, Pennsylvania
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Mt. Pleasant, South Carolina
  - Spartanburg, South Carolina
  - Jackson, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Victoria, Texas
  - Waco, Texas
  - Chesapeake, Virginia
  - Danville, Virginia
  - Richmond, Virginia
  - Suffolk, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
- Australia (4):
  - Camperdown, New South Wales
  - Woodville South, South Australia
  - Hobart, Tasmania
  - Shenton Park, Western Australia
- Canada (7):
  - Kelowna, British Columbia
  - Victoria, British Columbia
  - Halifax, Nova Scotia
  - London, Ontario
  - Mississauga, Ontario
  - Toronto, Ontario
  - Québec, Quebec
- New Zealand (3):
  - Grafton, Auckland
  - Tauranga, Bay of Plenty
  - Hamilton
- Poland (7):
  - Kutno, Lodz Province
  - Biatystok
  - Elblag
  - Gmina Końskie
  - Katowice
  - Krakow
  - Poznan
- Switzerland (2):
  - Lausanne, Vlaud
  - Fribourg

REFERENCES:
- [Derived] Topless R, Noorbaloochi S, Merriman TR, Singh JA. Change in serum urate level with urate-lowering therapy initiation associates in the immediate term with patient-reported outcomes in people with gout. Semin Arthritis Rheum. 2022 Oct;56:152057. doi: 10.1016/j.semarthrit.2022.152057. Epub 2022 Jun 29. PMID 35835008
- [Derived] Dalbeth N, Jones G, Terkeltaub R, Khanna D, Fung M, Baumgartner S, Perez-Ruiz F. Efficacy and safety during extended treatment of lesinurad in combination with febuxostat in patients with tophaceous gout: CRYSTAL extension study. Arthritis Res Ther. 2019 Jan 7;21(1):8. doi: 10.1186/s13075-018-1788-4. PMID 30616614
- [Derived] Dalbeth N, Jones G, Terkeltaub R, Khanna D, Kopicko J, Bhakta N, Adler S, Fung M, Storgard C, Baumgartner S, Perez-Ruiz F. Lesinurad, a Selective Uric Acid Reabsorption Inhibitor, in Combination With Febuxostat in Patients With Tophaceous Gout: Findings of a Phase III Clinical Trial. Arthritis Rheumatol. 2017 Sep;69(9):1903-1913. doi: 10.1002/art.40159. Epub 2017 Aug 4. PMID 28597604
- See also: Related Info — http://www.gouttrial.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 330 participants were randomized and 324 participants were included in the Intent-to-Treat (ITT) population (ie, 6 subjects were randomized but not treated).
Period: Overall Study
Arm/Group | Lesinurad 200 mg + Febuxostat | Lesinurad 400 mg + Febuxostat | Placebo + Febuxostat
Started | 106 | 109 | 109
Completed | 79 | 84 | 87
Not Completed | 27 | 25 | 22
Not completed — Adverse Event | 7 | 6 | 4
Not completed — Gout Flare | 0 | 3 | 1
Not completed — Protocol Violation | 11 | 10 | 9
Not completed — Lost to Follow-up | 5 | 1 | 5
Not completed — Withdrawal by Subject | 3 | 4 | 3
Not completed — Death | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lesinurad 200 mg + Febuxostat | Lesinurad 400 mg + Febuxostat | Placebo + Febuxostat | Total
Number analyzed (Participants) | 106 | 109 | 109 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (11.0) | 53.3 (11.2) | 54.6 (10.9) | 54.1 (11.0)
Age, Customized [Number; unit: Participants] — <65 Years, >=65 Years
  Participants
    <65 Years | 89 | 90 | 89 | 268
    >=65 Years | 17 | 19 | 20 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 2 | 15
  Male | 100 | 102 | 107 | 309
Region of Enrollment [Number; unit: Participants]
  Australia | 6 | 6 | 4 | 16
  Canada | 9 | 2 | 6 | 17
  New Zealand | 2 | 6 | 5 | 13
  Poland | 8 | 10 | 14 | 32
  Switzerland | 0 | 1 | 1 | 2
  United States | 81 | 84 | 79 | 244

OUTCOME MEASURES:

1. Primary Outcome: Subjects With a Serum Urate (sUA) Level That is < 5.0 mg/dL by Month 6
Description: Proportion of subjects with an sUA level that is < 5.0 mg/dL by Month 6
Time Frame: 6 months, analysis after all subjects complete 12 months
Population: Intent-to-Treat Population
Measure: Number; unit: Proportion of Subjects
Groups:
- Lesinurad 200 mg + Febuxostat 80 mg: lesinurad 200 mg once daily (qd) plus febuxostat 80 mg
- Lesinurad 400 mg + Febuxostat 80 mg: lesinurad 400 mg qd plus febuxostat 80 mg
- Placebo + Febuxostat 80 mg: placebo qd plus febuxostat 80 mg
Arm/Group | Lesinurad 200 mg + Febuxostat 80 mg | Lesinurad 400 mg + Febuxostat 80 mg | Placebo + Febuxostat 80 mg
Number analyzed (Participants) | 106 | 109 | 109
Proportion of Subjects | 0.566 | 0.761 | 0.468
Statistical Analysis 1: Comparison: Lesinurad 200 mg + Febuxostat 80 mg vs Placebo + Febuxostat 80 mg; Test type: Superiority or Other; p = 0.1298, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.10, 95% CI 2-sided [-0.03 to 0.23]
Statistical Analysis 2: Comparison: Lesinurad 400 mg + Febuxostat 80 mg vs Placebo + Febuxostat 80 mg; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.29, 95% CI 2-sided [0.17 to 0.42]

2. Secondary Outcome: Complete Resolution of at Least One Target Tophus
Description: Proportion of subjects who experience complete resolution of at least 1 target tophus by Month 12
Time Frame: 12 Months
Population: Intent-to-Treat Population
Measure: Number; unit: Proportion of Subjects
Arm/Group | Lesinurad 200 mg + Febuxostat 80 mg | Lesinurad 400 mg + Febuxostat 80 mg | Placebo + Febuxostat 80 mg
Number analyzed (Participants) | 106 | 109 | 109
Proportion of Subjects | 0.255 | 0.303 | 0.211
Statistical Analysis 1: Comparison: Lesinurad 200 mg + Febuxostat 80 mg vs Placebo + Febuxostat 80 mg; Test type: Superiority or Other; p = 0.4453, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.04, 95% CI 2-sided [-0.07 to 0.16]
Statistical Analysis 2: Comparison: Lesinurad 400 mg + Febuxostat 80 mg vs Placebo + Febuxostat 80 mg; Test type: Superiority or Other; p = 0.1149, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.09, 95% CI 2-sided [-0.02 to 0.21]

3. Secondary Outcome: Complete or Partial Response of at Least One Tophus
Description: Proportion of subjects with a best tophus response on at least 1 target tophus of complete (disappearance of at least 1 target tophus) or partial (≥ 50% decrease in the area of at least 1 target tophus) resolution by Month 12
Time Frame: 12 Months
Population: Intent-to-Treat Population
Measure: Number; unit: Proportion of Subjects
Arm/Group | Lesinurad 200 mg + Febuxostat 80 mg | Lesinurad 400 mg + Febuxostat 80 mg | Placebo + Febuxostat 80 mg
Number analyzed (Participants) | 106 | 109 | 109
Proportion of Subjects | 0.566 | 0.587 | 0.505
Statistical Analysis 1: Comparison: Lesinurad 200 mg + Febuxostat 80 mg vs Placebo + Febuxostat 80 mg; Test type: Superiority or Other; p = 0.6450, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.03, 95% CI 2-sided [-0.10 to 0.17]
Statistical Analysis 2: Comparison: Lesinurad 400 mg + Febuxostat 80 mg vs Placebo + Febuxostat 80 mg; Test type: Superiority or Other; p = 0.4118, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.06, 95% CI 2-sided [-0.08 to 0.19]

4. Secondary Outcome: Quality of Life
Description: Proportion of subjects with an improvement from Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) of at least 0.25 at Month 12. The HAQ-DI assesses a patient's level of functional ability with items scores ranging from 0-3 with 0 being the least disability.
Time Frame: 12 Months
Population: Intent-to-Treat Population
Measure: Number; unit: Proportion of Subjects
Arm/Group | Lesinurad 200 mg + Febuxostat 80 mg | Lesinurad 400 mg + Febuxostat 80 mg | Placebo + Febuxostat 80 mg
Number analyzed (Participants) | 77 | 78 | 80
Proportion of Subjects | 0.442 | 0.333 | 0.525
Statistical Analysis 1: Comparison: Lesinurad 200 mg + Febuxostat 80 mg vs Placebo + Febuxostat 80 mg; Test type: Superiority or Other; p = 0.3034, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.08, 95% CI 2-sided [-0.24 to 0.07]
Statistical Analysis 2: Comparison: Lesinurad 400 mg + Febuxostat 80 mg vs Placebo + Febuxostat 80 mg; Test type: Superiority or Other; p = 0.0210, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.19, 95% CI 2-sided [-0.34 to -0.04]

ADVERSE EVENTS:
Arm/Group | Lesinurad 200 mg + Febuxostat | Lesinurad 400 mg + Febuxostat | Placebo + Febuxostat
Serious Adverse Events (participants affected / at risk) | 6/106 | 9/109 | 10/109
Other Adverse Events (participants affected / at risk) | 50/106 | 59/109 | 34/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lesinurad 200 mg + Febuxostat (N=106) | Lesinurad 400 mg + Febuxostat (N=109) | Placebo + Febuxostat (N=109)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.02% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lesinurad 200 mg + Febuxostat (N=106) | Lesinurad 400 mg + Febuxostat (N=109) | Placebo + Febuxostat (N=109)
Dental caries (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (4) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 7 (7) | 4 (4)
Influenza (Infections and infestations) | 6 (6) | 2 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 10 (10) | 15 (15) | 9 (12)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 7 (9) | 3 (3)
Excoriation (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 4 (4) | 6 (6) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 8 (12) | 4 (5)
Blood creatine phosphokinase increased (Investigations) | 6 (8) | 4 (4) | 3 (3)
Blood creatinine increased (Investigations) | 7 (7) | 8 (11) | 3 (3)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 6 (7) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (9) | 9 (9) | 4 (4)
Headache (Nervous system disorders) | 10 (11) | 6 (7) | 8 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (9) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 12 (13) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.